CLINICAL TRIAL: NCT01711307
Title: Operative vs. Non-Operative Treatment of Acute Ruptures of the Achilles Tendon: A Multi-centered Randomized Control Trial Using Standardized Objective and Subjective Outcome Measurement to Determine Rerupture Rate.
Brief Title: Operative vs. Non-Operative Treatment of Acute Ruptures of the Achilles Tendon
Acronym: AchillesRCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Glazebrook (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Mark Glazebrook, Dr Mark Glazebrook, MSc,PHD, Dip Sports Med, MD FRCS(c), Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version1
Record Dates: First submitted 2012-10-11; First posted 2012-10-22 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Ruptured Achilles Tendon
Keywords: Achilles; Rupture
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-operative (Experimental): cast applied within 48 hours
  Interventions: Procedure: non-operative
- operative (Active Comparator): cast applied within 48 hours and surgery within 14 days
  Interventions: Procedure: operative

INTERVENTIONS:
Procedure: operative
  Arms: operative
Procedure: non-operative — casting within 48 hrs
  Arms: non-operative

SUMMARY:
The proposed trial is a multi-centre prospective randomized controlled trial comparing outcomes of patients with acute Achilles tendon ruptures treated either non-operatively or with open operative tendon repair. All patients will undergo accelerated functional rehabilitation. The primary outcome measure is Achilles tendon re-rupture rate.

DETAILED DESCRIPTION:
Equivalent clinical outcomes to surgical repair; reduced morbidity and disability to subjects through elimination of a surgical repair; reduction of cost to patients by eliminating need for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Complete mid-substance rupture of the Achilles tendon as diagnosed on clinical exam
* Present for initial assessment and treatment with application of a plantar-flexed cast within 48 hours of their injury.
* Referred to one of the participating orthopaedics surgeons in a timely fashion so as to allow for further treatment (operative repair or initiation of the rehabilitation protocol) within 14 days of their injury.

Exclusion Criteria:

* Open Achilles injury
* Achilles injury that is not a mid-substance tendon injury
* Any additional injury to the ipsilateral lower extremity
* Contraindication to surgery or anesthetic
* (Physical or mental) that may interfere with compliance with the rehabilitation protocol
* Any known factor for increased risk of Achilles tendon rupture (i.e. diabetes mellitus, immunosuppressive therapy including local or systemic steroids, and fluoroquinolone use).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2012-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Operative vs non operative Treatment of acute ruptures of Achilles tendon. | 1 year
  The primary outcome measure is Achilles tendon re-rupture rate

SECONDARY OUTCOMES:
Operative vs. Non-Operative Treatment of Acute Ruptures of the Achilles Tendon | 2 year
  1. The Achilles tendon Total Rupture Score (ATRS)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mark Glazebrook, MD, Principal Investigator — Capital Health District Authority
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
COA AAOS AOFAS